CLINICAL TRIAL: NCT01041131
Title: Laparoscopic Revisional Gastric Bypass Surgery for Failed and/or Complicated Open Vertical Banded Gastroplasty: Our Experience With 70 Patients
Brief Title: Laparoscopic Revision of Vertical Banded Gastroplasty to Gastric Bypass
Acronym: VBG
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2009073; U1111-1113-0085 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-31 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Clinically Severe Obesity; Inadequate Weight Loss; Obesity Recidivism
Keywords: Obesity; Obesity recidivism; Inadequate Initial Weight Loss; Technical bariatric complications; Complicated gastroplasty; Failed gastroplasty; Gastroesophageal reflux disease; Revisional gastric bypass; Conversion bariatric surgery; Re-operative bariatric surgery; Technical complications of vertical gastroplasty; Complicated vertical gastroplasty
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Failed and/or Complicated VBG

SUMMARY:
The main aim of this study is to analyze and report the intermediate term outcomes after laparoscopic revision Roux-en-Y gastric bypass (RYGB) surgery for failed and/or complicated Vertical Banded Gastroplasty (VBG). The foremost outcome measurements are 1) Fat loss mainly measured as weight loss and expressed as trends in BMI, %EWL, and/or %EBL. 2) Trend in Comorbidity status. 3) Subjective Satisfaction and Health-Related Quality of Life "HR-QoL" are measured by a standardized, non-validated satisfaction questionnaire and by a validated, disease-specific worldwide used HR-QoL questionnaire. 4) Morbidity & Mortality include nutritional status and metabolic complications.

Consequently, secondary objectives of this study are the following. 1) To assess failure rate defined as percentage of excess weight loss < 50%, lowest BMI >35 for morbidly obese (MO) or >40 for superobese (SO), and/or lack of resolution/improvement of major comorbidities at the point in time when assessed at each postoperative year after the surgery under study. 2) To evaluate the metabolic and nutritional status by measurements of particular clinical and biochemical parameters.

DETAILED DESCRIPTION:
There is no real standardization for any of the previously stated "modern standard bariatric procedures" endorse by the ASMBS; thus, outcomes vary widely with each one of them. For purposes of this study, the term Vertical Banded Gastroplasty (VBG) is used to encompass several types of vertical gastroplasties with a reinforced stoma such as nondivided vertical banded gastroplasty, nondivided vertical ringed gastroplasty, transected or divided vertical ringed or banded gastroplasties among others. VBG, in various forms, was used extensively for more than 2 decades after its original description by Mason in 198217. Designed to avoid the long-term nutritional implications and complexity of gastric bypass, VBG evolved and permitted us to infer some mechanism of failure and modify other bariatric procedures. Regardless of a laparoscopic approach, VBG is no longer a viable option for the treatment of morbid obesity because of less overall weight loss, high failure and late complication rates.

The following are the main investigators that have addressed diverse revisional strategies including restoration or conversion of VBG into a modern bariatric procedure, either by open or laparoscopic approach, because of failure and/or technical complications:

I. Open approach. Most of the scientific literature available on redo bariatric surgery is based on open surgery series. There is no consensus on what type of revisional procedure is the best; however, there are several options available.

A) Restoration or re-VBG is no longer a viable option.

1. In a study of 122 gastroplasties, Sugerman et al reported that four out of ten re-VBG patients required a third revision.
2. With a Kaplan-Meyer analysis, Van Gemert et al found that re-VBG carry a secondary revisional rate of 68% over a 5-year period vs. a 0% rate after conversion to RYGB.

B) Other revisional option is adjustable gastric band (AGB).

1. In 2001, Charuzi et al described revisional adjustable gastric band after diverse failed primary bariatric procedures. However, they reported their compound outcome results without subset analysis.
2. In the same year, Taskin et al published a series of 7 patients undergoing revisional adjustable gastric banding and obtained comparable results with primary AGB at 2 years. However, all patients had preoperatively identified a staple-line failure and the morbi-mortality was not stated.
3. In 2004, Gavert et al analyzed 47 patients undergoing laparoscopic revisional surgery using AGB with a mean BMI at 16 months of 32 and an early complication rate of 4%. No mortality was reported.

C) Other recently added strategy to the revisional armamentarium is Sleeve Gastrectomy (SG). Iannelli et al in 2009 published the analysis of 41 patients undergoing revisional SG for failed AGB (n=36) or VBG (n=5). No subset analysis was provided however postoperative morbidity was 12.2%; at a mean of 13.4 months, mean BMI, %EWL, and %EBL were 42.7%, 42.7%, 47.4% respectively; and re-operation rate for failure was 14.6% (n=6).

D) Another reported revisional procedure is Biliopancreatic Diversion with Duodenal Switch (BPD-DS).

1) Of 47 patients revised to BPD-DS by Keshishian et al, 16 had a VBG as the primary bariatric procedure. Their reported outcome data is mixed with failed RYGB (n=31). Although this revisional strategy carried a higher major morbidity rate (12.8%), the weight loss was comparable to the primary BPD-DS.

E) However, most published studies about revisional surgery for failed or complicated VBG support RYGB as a revisional procedure. Previously some investigators have shown the RYGB superiority over VBG. Specifically, RYGB has more overall weight loss, less late complications and less revision rates than VBG.

1. Sugerman and van Gemert have compared restoration vs. conversion to RYGB, highlighting again the supremacy of RYGB, mostly based on the revisional rate and weight loss. Therefore, conversion of VBG to RYGB seems to be logical.
2. In 1993, Sapala et al (n=20) reported technical strategies for converting VBG to RYGB. Major early morbidity occurred in 4 patients (20%).
3. In 1996, Sugerman et al (n=53) obtained a statistical significant increased of %EWL from 36% to 67% and 20% to 70% in "big eaters" and in "sweets eaters", respectively. Weight loss for revisional RYGB was comparable to the one after primary RYGB. Upper GI symptoms were completely resolved. Morbidity was described in 26 patients (49%).
4. In 1998, Capella & Capella (n=60), with an adjusted Roux-limb length for BMI, reported at 1 year follow-up 68% and 76% EWL for proximal and distal RYGB patients, respectively.
5. In 2004, Cordera et al (n=54), with an adjusted Roux-limb length for BMI, reported weight loss as a decrease in BMI from 46 Kg/m2, at the time of conversion, to 35 Kg/m2 at 6.1 years (94% patients). In addition, comorbidities status measured by medication consumption were ameliorated and subjective patient satisfaction at survey was high (90%). However, one year post-conversion 41% of the series had a BMI greater than 35 Kg/m2.
6. In 2005, Gonzalez et al (n=28), on a 5 basic steps of standardized technique and adjusted Roux-limb length for BMI, reported a decrease in BMI from 40 Kg/m2 to 32 Kg/m2 at 16 months of follow-up. Overall %EWL was 48% (range, 3-71%), however, resolution in comorbidities ranged from 50 to 86%. Early morbidity occurred in 9 patients (32%).
7. In 2007, van Dielen et al (n=41) revised 11 AGB and 30 VBG most of them by open approach. BMI decreased from 37.7 to 29.4 at 12 months while %EWL increased from 39.1% to 75.4% (p< 0.001). Major early (n=4) and late (n=10) complications were registered. No remission in comorbidities was observed35.
8. In the 2007 outcome analysis by Schouten et al (n=101) found out that the effect on weight is dependent of the indication for revision. Weight recidivism patient's BMI decreased from 40.5 Kg/m2 to 30.1 Kg/m2; excessive weight loss patients BMI increased from 22.3 Kg/m2 to 25.3 Kg/m2; and adequate response patients to VBG but with severe eating difficulties remained stable (29.8 Kg/m2 to 29.0 Kg/m2) all after a mean follow-up of 38 months.

Therefore, based on all this observational studies, the open conversion of VBG to RYGB has been demonstrated to be an effective procedure with defined complications.

II. Laparoscopic Approach. Increasing experience with minimally invasive bariatric surgery has prompted surgeons to approach most revisions procedures laparoscopically.

A) Because most published studies about open revisional surgery for failed and/or complicated VBG support RYGB as the revisional procedure of choice, most laparoscopic bariatric surgeons follow this principle.

1. Csepel et al (n=7), in 2001, reported their initial experience with laparoscopic approach for revision bariatric surgery; 6 patients in this group had failed VBG. Pre-revisional BMI decreased from 42.2 to 37.2 without specifying the length of follow-up or resolution of comorbidities. Three major complications (42.8%) were reported.
2. Gagner et al reported their continued revisional experience with 12 patients, a subgroup of 27, who underwent reoperation for failed VBG. Overall, pre-revisional BMI decreased from 42.7 Kg/m2 to 35.9 Kg/m2 after 8 months of follow-up (p< 0.001) with a 22% complication rate. Resolution of comorbidities was not stated.
3. Gagne et al, in 2005, reported their experience revising laparoscopically 25 patients with a 24% morbidity rate, 51 %EWL at 3 years, 100% resolution of diabetes and 63% resolution of hypertension.
4. In 2005, Calmes et al (n=49) reported their initial experience with laparoscopic revisional RYGB with 15 patients, a subset of 49, who had a failed or complicated VBG. Overall complication rate of 36% (Major 4%, minor 20% and late 14%) 70-75% of the patients at 4 years had a BMI less than 35.
5. In 2007, Suter et al reported their accumulative experience with open (n=47) and laparoscopic (n=74) revisional RYGB. The primary procedures were LAGB (n=82), VBG (36) and RYGB (n=3). Overall morbidity was 26.4% and 75% of the patients at 5 years had a BMI less than 35 Kg/m2.
6. Van Dessel et al, in 2008, published his experience on 36 patients with laparoscopic revisional RYGB for failed restrictive procedures ( 14 VBG, 20 AGB, and 2 SG). After a short follow-up of 6.6 months, early and late morbidity was 30% and 16.7%, respectively; BMI dropped from 38.8 kg/m2 to 30.9 kg/m2; and a higher but not significant early morbidity rate for the complicated vs. the failed subgroups

Summarizing, there is lack of standardization of primary and revisional bariatric surgery compounded by a scant long-term outcome data. The treatment of inadequate weight loss, weight recidivism, and most severe technical complications after primary bariatric surgery remains refractory to non-operative treatment. Failure and secondary revisional rates after VBG can be as high as 56% and 68%, respectively. Indication for further surgical intervention remains controversial, as does what type of procedure to recommend but the most widely documented and with best risk-benefit ratio option is RYGB. After extensive literature search, there is no outcome study employing a laparoscopic revisional strategy with a HSA reporting outcomes comparable to primary gastric bypass in an unselected obese population. Thus, we formally analyze our experience with the laparoscopic approach to these complex and challenging patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients status post failed and/or complicated VBG undergoing laparoscopic revisional RYGB

Exclusion Criteria:

* Patients with prior major conversion, revision, and/or esophago-gastric surgery
* Conversion performed by open approach
* Conversion performed somewhere else with follow-up by our program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients status post failed and/or complicated Vertical Banded Gastroplasty (VBG) undergoing conversion to laparoscopic Roux-en-Y gastric bypass (RYGB)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | at discharge, 1 week, 3 weeks, 8 weeks, 3 months, 6 months, 1 year and annually thereafter for up to 8 years
Weight loss expressed as Body Mass Index and Percentage excess weight loss | at 6 months, 1 year and annually thereafter for up to 8 years
Remission or improvement of symptoms | at 6 months, 1 year and annually thereafter for up to 8 years

SECONDARY OUTCOMES:
Length of operative time which is defined as the time duration of operation measured in minutes from the first skin incision to the final closure of the skin incision | It is measured in minutes from the first skin incision to the final closure of the skin incision at the time of revisional surgery under study. It is a transoperative measure of outcome of the surgery under study
Remission or improvement of comorbidities | at 6 months, 1 year, and annually thereafter for up to 8 years
Length of Hospital Stay which is a measured of surgical recovery quantified and reported in days. It is a hospital pre-discharge traditional measure of outcome. | It is measured in days from the admission date to the discharge date for the hospitalization pertaining to revisional surgery under study.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] ASMBS www.asbs.org/htm/Private/resolution.html
- [Background] O'Brien PE, McPhail T, Chaston TB, Dixon JB. Systematic review of medium-term weight loss after bariatric operations. Obes Surg. 2006 Aug;16(8):1032-40. doi: 10.1381/096089206778026316. PMID 16901357
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- [Background] Mason EE. Vertical banded gastroplasty for obesity. Arch Surg. 1982 May;117(5):701-6. doi: 10.1001/archsurg.1982.01380290147026. PMID 7073493
- [Background] Sugerman HJ, Wolper JL. Failed gastroplasty for morbid obesity. Revised gastroplasty versus Roux-Y gastric bypass. Am J Surg. 1984 Sep;148(3):331-6. doi: 10.1016/0002-9610(84)90465-3. PMID 6383098
- [Background] van Gemert WG, van Wersch MM, Greve JW, Soeters PB. Revisional surgery after failed vertical banded gastroplasty: restoration of vertical banded gastroplasty or conversion to gastric bypass. Obes Surg. 1998 Feb;8(1):21-8. doi: 10.1381/096089298765555006. PMID 9562482
- [Background] Kyzer S, Raziel A, Landau O, Matz A, Charuzi I. Use of adjustable silicone gastric banding for revision of failed gastric bariatric operations. Obes Surg. 2001 Feb;11(1):66-9. doi: 10.1381/096089201321454132. PMID 11361171
- [Background] Taskin M, Zengin K, Unal E, Sakoglu N. Conversion of failed vertical banded gastroplasty to open adjustable gastric banding. Obes Surg. 2001 Dec;11(6):731-4. doi: 10.1381/09608920160558678. PMID 11775571
- [Background] Gavert N, Szold A, Abu-Abeid S. Safety and feasibility of revisional laparoscopic surgery for morbid obesity: conversion of open silastic vertical banded gastroplasty to laparoscopic adjustable gastric banding. Surg Endosc. 2004 Feb;18(2):203-6. doi: 10.1007/s00464-002-8643-y. Epub 2003 Nov 21. PMID 14625748
- [Background] Iannelli A, Schneck AS, Ragot E, Liagre A, Anduze Y, Msika S, Gugenheim J. Laparoscopic sleeve gastrectomy as revisional procedure for failed gastric banding and vertical banded gastroplasty. Obes Surg. 2009 Sep;19(9):1216-20. doi: 10.1007/s11695-009-9903-x. Epub 2009 Jun 27. PMID 19562420
- [Background] Keshishian A, Zahriya K, Hartoonian T, Ayagian C. Duodenal switch is a safe operation for patients who have failed other bariatric operations. Obes Surg. 2004 Oct;14(9):1187-92. doi: 10.1381/0960892042387066. PMID 15527632
- [Background] Sugerman HJ, Starkey JV, Birkenhauer R. A randomized prospective trial of gastric bypass versus vertical banded gastroplasty for morbid obesity and their effects on sweets versus non-sweets eaters. Ann Surg. 1987 Jun;205(6):613-24. doi: 10.1097/00000658-198706000-00002. PMID 3296971
- [Background] Sugerman HJ, Londrey GL, Kellum JM, Wolf L, Liszka T, Engle KM, Birkenhauer R, Starkey JV. Weight loss with vertical banded gastroplasty and Roux-Y gastric bypass for morbid obesity with selective versus random assignment. Am J Surg. 1989 Jan;157(1):93-102. doi: 10.1016/0002-9610(89)90427-3. PMID 2910132
- [Background] Hall JC, Watts JM, O'Brien PE, Dunstan RE, Walsh JF, Slavotinek AH, Elmslie RG. Gastric surgery for morbid obesity. The Adelaide Study. Ann Surg. 1990 Apr;211(4):419-27. doi: 10.1097/00000658-199004000-00007. PMID 2181950
- [Background] Fobi MA. Vertical Banded Gastroplasty vs Gastric Bypass: 10 years follow-up. Obes Surg. 1993 May;3(2):161-164. doi: 10.1381/096089293765559511. PMID 10757913
- [Background] Sapala JA, Bolar RJ, Bell JP, Sapala MA. Technical Strategies for Converting the Failed Vertical Banded Gastroplasty to the Roux-en-Y Gastric Bypass. Obes Surg. 1993 Nov;3(4):400-409. doi: 10.1381/096089293765559115. PMID 10757953
- [Background] Sugerman HJ, Kellum JM Jr, DeMaria EJ, Reines HD. Conversion of failed or complicated vertical banded gastroplasty to gastric bypass in morbid obesity. Am J Surg. 1996 Feb;171(2):263-9. doi: 10.1016/S0002-9610(97)89565-7. PMID 8619465
- [Background] Capella RF, Capella JF. Converting vertical banded gastroplasty to a lesser curvature gastric bypass: technical considerations. Obes Surg. 1998 Apr;8(2):218-24. doi: 10.1381/096089298765554854. PMID 9730398
- [Background] Cordera F, Mai JL, Thompson GB, Sarr MG. Unsatisfactory weight loss after vertical banded gastroplasty: is conversion to Roux-en-Y gastric bypass successful? Surgery. 2004 Oct;136(4):731-7. doi: 10.1016/j.surg.2004.05.055. PMID 15467656
- [Background] Gonzalez R, Gallagher SF, Haines K, Murr MM. Operative technique for converting a failed vertical banded gastroplasty to Roux-en-Y gastric bypass. J Am Coll Surg. 2005 Sep;201(3):366-74. doi: 10.1016/j.jamcollsurg.2005.04.022. PMID 16125069
- [Background] Van Dielen FM, Stevens D, Zoete JP, et al. Results after gastric bypass as revisional surgery. Obes Surg 2007;17:1055.
- [Background] Schouten R, van Dielen FM, van Gemert WG, Greve JW. Conversion of vertical banded gastroplasty to Roux-en-Y gastric bypass results in restoration of the positive effect on weight loss and co-morbidities: evaluation of 101 patients. Obes Surg. 2007 May;17(5):622-30. doi: 10.1007/s11695-007-9106-2. PMID 17658021
- [Background] de Csepel J, Nahouraii R, Gagner M. Laparoscopic gastric bypass as a reoperative bariatric surgery for failed open restrictive procedures. Surg Endosc. 2001 Apr;15(4):393-7. doi: 10.1007/s004640000347. Epub 2001 Feb 6. PMID 11395822
- [Background] Gagner M, Gentileschi P, de Csepel J, Kini S, Patterson E, Inabnet WB, Herron D, Pomp A. Laparoscopic reoperative bariatric surgery: experience from 27 consecutive patients. Obes Surg. 2002 Apr;12(2):254-60. doi: 10.1381/096089202762552737. PMID 11975224
- [Background] Gagne DJ, Goitein D, Papasavas PK, et al. Laparoscopic revision of vertical banded gastroplasty to Roux-en-Y gastric bypass: an outcome analysis. Obes Surg 2005;1:243.
- [Background] Calmes JM, Giusti V, Suter M. Reoperative laparoscopic Roux-en-Y gastric bypass: an experience with 49 cases. Obes Surg. 2005 Mar;15(3):316-22. doi: 10.1381/0960892053576785. PMID 15826463
- [Background] Suter M, Calmes JM, Paroz A, et al. Revisional Roux-en-Y gastric bypass: 8-year experience with 121 patients. Obes Sug 2007;17:1057.
- [Background] Van Dessel E, Hubens G, Ruppert M, Balliu L, Weyler J, Vaneerdeweg W. Roux-en-Y gastric bypass as a re-do procedure for failed restricive gastric surgery. Surg Endosc. 2008 Apr;22(4):1014-8. doi: 10.1007/s00464-007-9576-2. Epub 2007 Oct 18. PMID 17943380
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/